CLINICAL TRIAL: NCT02886286
Title: Randomized, Double Blind, Cross Over Study Comparing Effectiveness of Traditional Opioids Versus Opioids in Admixture With Bupivacaine Upon Self-administration of Boluses Via a Personal Therapy Manager (PTM) in Intrathecal Pumps
Brief Title: Patient Controlled Intrathecal Analgesia With Bupivacaine for Chronic Low Back Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Salim M Hayek, MD, PhD, Chief, Division of Pain Medicine, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2-16-24
Record Dates: First submitted 2016-08-18; First posted 2016-09-01 (Estimated); Results first posted 2022-03-24 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-02

CONDITIONS: Pain, Intractable; Breakthrough Pain; Chronic Pain
MeSH Terms: conditions — Pain, Intractable; Breakthrough Pain; Chronic Pain | interventions — Bupivacaine; Analgesics, Opioid; Fentanyl; Hydromorphone; Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bupivacaine + Opioid (Experimental): Intrathecal solution has bupivacaine with an opioid (hydromorphone, fentanyl or morphine). Patients will administer PTM bolus of bupivacaine with opioid. The bolus will be administered over 2 minutes and will have a variable frequency depending on patient's need but the number of boluses should be >2 and <10. The bupivacaine dosage would range between 0.4 and 1.5 mg per bolus. The opioid dose will vary depending on the concentration of the opioid in the solution.
  Interventions: Drug: Bupivacaine; Drug: Opioid
- Opioid (Active Comparator): Intrathecal solution has only an opioid (hydromorphone, fentanyl or morphine) and no bupivacaine. Patients will administer PTM bolus of opioid without bupivacaine. This opioid bolus dose would be the same as they would have received prior to enrolling in the study (with bupivacaine). The bolus will be administered over 2 minutes and will have a variable frequency depending on patient's need but the number of boluses should be >2 and <10.
  Interventions: Drug: Opioid

INTERVENTIONS:
Drug: Bupivacaine — Patient-activated intrathecal bolus for incident pain
  Arms: Bupivacaine + Opioid
Drug: Opioid — Patient-activated intrathecal bolus for incident pain
  Other Names: Fentanyl; Hydromorphone; Morphine

SUMMARY:
The purpose of this study is to determine whether the local anesthetic bupivacaine delivered intrathecally in small doses via PTM self-administered boluses significantly improves the breakthrough pain and functional status of patients with chronic intractable pain who are managed with an intrathecal drug delivery system.

DETAILED DESCRIPTION:
Methodology /Technical Approach:

Seventeen patients who are already using SynchroMed II pump containing an admixture of bupivacaine and an opioid and using PTM doses will receive Solution A during the first week of the study and will be crossed over to Solution B during the second week of the study. Solution A and Solution B would consist of either the patient's usual intrathecal opioid with bupivacaine at the same concentrations or the usual patient's intrathecal opioid at the same concentration but without bupivacaine. Only the Investigational Pharmacy at University Hospitals Case Medical Center (UHCMC) would be aware of the contents of Solution A and Solution B. Patients and study personnel in the Pain Medicine Division would be blinded to the solution content. The sequence of pump refills will be as follows:

* Week I: Patients will have the intrathecal pumps refilled with 10 milliliters of a Solution A or B, after removal of residual volume of baseline solution.
* Week II: IT pump will be filled with 10 ml of Solution A or B (whichever solution subject did not receive Week 1), after removal of residual volume from Week I.

Both patients and the evaluating physician will be blinded. In order to accomplish this, only the central compounding (investigational) pharmacy at UHCMC would make two solutions labeled: A or B respectively. Study subjects will be randomized and randomization order will be held at the pharmacy that will supply the medication. Patients will be kept on each solution for one week. Data will be collected daily

Primary outcome measures will include 0-10 numerical rating scale (NRS) or Visual Analogue Scale (VAS) both immediately before and within 30 minutes after a PTM bolus. Patients will be provided with a diary to record pain scores just before a PTM bolus and the lowest pain score within half an hour after a PTM bolus. Only 5 recording per day on days 3-7 and 10-14 will be available on the diary-thus patients would record pain scores only before and after the first 5 PTM boluses. Only the scores before and after the first 3 successful PTM boluses would be considered. Successful PTM activations would be determined by review of the patient PTM diary and the internal log from the intrathecal drug delivery system. Each recording on the PTM diary would be time matched to the successful PTM activation code in the internal log. This will obviate any potential mis-administered bolus whereby the patient does not activate the bolus device appropriately. Secondary outcome measures will include average NRS pain scores for the week, functional capacity as evaluated by the Oswestry disability index (ODI) scores, Global Impression of Change and painDETECT. Other relevant data such as number of boluses used and paresthetic sensation post bolus (if felt)/patient guess of blinding arm would be recorded.

ELIGIBILITY:
Inclusion Criteria

* Age more than 30 years implanted with an intrathecal drug delivery device.
* Intrathecal pump patients on stable dose for the last 3 months.
* Using on average more than 2 and less than 10 PTM doses per day
* Intrathecal medication admixture consisting of bupivacaine and another opioid (fentanyl or hydromorphone or morphine)

Exclusion Criteria

* Using 10 or more PTM bolus doses per day or 2 or less PTM bolus doses per day
* Pending litigation or worker compensation claim
* Any recent (less than 3 month) procedures in spine (surgeries) or catheter adjustments.
* Recent pump dose adjustment within the past 3 months
* Pumps with medications other than bupivacaine/opioid combination.
* Pregnant or breast feeding

Ages: 31 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2016-05; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Case Medical Center, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Bupivacaine + Opioid First, Then Opioid: Intrathecal solution has bupivacaine with an opioid (hydromorphone, fentanyl or morphine). Patients will administer PTM bolus of bupivacaine with opioid. The bolus will be administered over 2 minutes and will have a variable frequency depending on patient's need but the number of boluses should be >2 and <10. The bupivacaine dosage would range between 0.4 and 1.5 mg per bolus. The opioid dose will vary depending on the concentration of the opioid in the solution.
  Bupivacaine: Patient-activated intrathecal bolus for incident pain
  Opioid: Patient-activated intrathecal bolus for incident pain
  Patients received Bupivacaine + Opioid first for 7 days. Patients were crossed over at day 8 to receive Opioid only. Bolus delivery was locked out after each medication change for one to two days. Data were collected on days 4-7 and days 11-14.
- Opioid First, Then Bupivacaine + Opioid: Intrathecal solution has only an opioid (hydromorphone, fentanyl or morphine) and no bupivacaine. Patients will administer PTM bolus of opioid without bupivacaine. This opioid bolus dose would be the same as they would have received prior to enrolling in the study (with bupivacaine). The bolus will be administered over 2 minutes and will have a variable frequency depending on patient's need but the number of boluses should be >2 and <10.
  Opioid: Patient-activated intrathecal bolus for incident pain
  Patients received Opioid only first for 7 days. Patients were crossed over at day 8 to receive Bupivacaine + Opioid. Bolus delivery was locked out after each medication change for one to two days. Data were collected on days 4-7 and days 11-14.
Period: Overall Study
Arm/Group | Bupivacaine + Opioid First, Then Opioid | Opioid First, Then Bupivacaine + Opioid
Started | 8 | 9
Completed (one patient had an unrelated motor stall of the pump) | 8 | 8
Not Completed | 0 | 1
Not completed — pump motor stall | 0 | 1

BASELINE CHARACTERISTICS:
Population: Participants who finished study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Bupivacaine + Opioid | Opioid | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 4 | 8
  >=65 years | 4 | 4 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.125 (8.96) | 63.75 (10.8) | 63.43 (9.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 3 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 7 | 8 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 16

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Numerical Rating Pain Scale (NRS)
Description: Patients will be provided with a diary to record pain scores just before a PTM bolus and the lowest pain score within half an hour after a PTM bolus.
  Numerical Rating Pain Scale (NRS): scale from 0-10 0 = no pain 10 = worst imaginable pain
Time Frame: Before self-administered bolus using Patient Therapy Manager device (PTM) and within 30 minutes of PTM bolus
Population: All participants who received each intervention were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Bupivacaine + Opioid: Intrathecal solution has bupivacaine with an opioid (hydromorphone, fentanyl or morphine). Patients will administer PTM bolus of bupivacaine with opioid. The bolus will be administered over 2 minutes and will have a variable frequency depending on patient's need but the number of boluses should be >2 and <10. The bupivacaine dosage would range between 0.4 and 1.5 mg per bolus. The opioid dose will vary depending on the concentration of the opioid in the solution.
  Bupivacaine: Patient-activated intrathecal bolus for incident pain
  Opioid: Patient-activated intrathecal bolus for incident pain
  Patients who received Bupivacaine + Opioid for 7 days, either in the first 7 days or last 7 days of the study. Bolus delivery was locked out after each medication change for one to two days. Data were collected on days 4-7 and days 11-14.
- Opioid: Intrathecal solution has only an opioid (hydromorphone, fentanyl or morphine) and no bupivacaine. Patients will administer PTM bolus of opioid without bupivacaine. This opioid bolus dose would be the same as they would have received prior to enrolling in the study (with bupivacaine). The bolus will be administered over 2 minutes and will have a variable frequency depending on patient's need but the number of boluses should be >2 and <10.
  Opioid: Patient-activated intrathecal bolus for incident pain
  Patients received Opioid only for 7 days, either in the first 7 days or last 7 days of the study. Bolus delivery was locked out after each medication change for one to two days. Data were collected on days 4-7 and days 11-14.
Arm/Group | Bupivacaine + Opioid | Opioid
Number analyzed (Participants) | 16 | 16
units on a scale | 1.87 (1.4) | 1.81 (1.47)

2. Secondary Outcome: Change From Baseline in Oswestry Disability Index (ODI)
Description: Oswestry Disability Index (ODI): calculated as a percentage based on scores from 0-5 in 10 categories (pain intensity, personal care, lifting, walking, sitting, standing, sleeping, sex life, social life, travelling). 0 signifies no pain interference while 5 signifies maximum possible pain interference in the 10 categories. Scores from 0-5 for 10 categories are added and divided by total possible score (50) X 100 to give percentage.
  Interpretation of percentage scores:
  0 - 20% minimal disability 21-40% moderate disability 41-60% severe disability 61-80% crippled 81-100% either bed bound or patient is exaggerating symptoms
Time Frame: Day 0, 7, 14, score at day 7 or day 14 reported
Population: All participants who received each intervention were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bupivacaine + Opioid | Opioid
Number analyzed (Participants) | 16 | 16
units on a scale | .88 (9.4) | 2.67 (9.02)

3. Secondary Outcome: Change From Baseline in Patient Global Impression of Change (PGIC)
Description: Patient Global Impression of Change (PGIC): reflects patient's belief about the efficacy of treatment
  1. = very much improved
  2. = much improved
  3. = minimally improved
  4. = no change
  5. = worse
  6. = much worse
  7. = very much worse
Time Frame: Day 0, 7, 14, score at day 7 or day 14 reported
Population: All participants who received each intervention were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bupivacaine + Opioid | Opioid
Number analyzed (Participants) | 16 | 16
units on a scale | -0.06 (2.11) | 1.25 (1.81)

4. Secondary Outcome: Change From Baseline in painDETECT
Description: painDETECT is a nine-item questionnaire that consists of seven sensory symptom items for pain that are graded from 0= never to 5= strongly, one temporal item on pain-course pattern graded -1 to +1, and one spatial item on pain radiation graded 0 for no radiation or +2 for radiating pain. A total score that ranges from -1 to 38 can be calculated from the nine items, with higher scores indicating higher levels of pain.
Time Frame: Day 0, 7, 14, score at day 7 or day 14 reported
Population: All participants who received each intervention were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bupivacaine + Opioid | Opioid
Number analyzed (Participants) | 16 | 16
units on a scale | 0.69 (2.96) | 0.25 (4.75)

5. Secondary Outcome: Change From Baseline in Average Weekly Numeric Pain Rating Score (NRS)
Description: Average Weekly Numeric Pain Rating Score (NRS) over the past week
  Numerical Rating Pain Scale (NRS): scale from 0-10 0 = no pain 10 = worst imaginable pain
Time Frame: Day 0, 7, 14, score at day 7 or day 14 reported
Population: All participants who received each intervention were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bupivacaine + Opioid | Opioid
Number analyzed (Participants) | 16 | 16
units on a scale | -0.47 (1.59) | -0.38 (1.69)

6. Secondary Outcome: Change From Baseline in Treatment Satisfaction
Description: A 5-point qualitative Likert scale was used to report measures of patient satisfaction (i.e., not satisfied at all, not satisfied, somewhat, satisfied, very satisfied). To quantify satisfaction, these responses were transformed to a scale of 0-4, with higher numbers representing greater levels of satisfaction.
Time Frame: Day 0, 7, 14, score at day 7 or day 14 reported
Population: All participants who received each intervention were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bupivacaine + Opioid | Opioid
Number analyzed (Participants) | 16 | 16
units on a scale | 2.36 (1.22) | 1.94 (1.18)

ADVERSE EVENTS:
Time Frame: 2 weeks
Description: Removing the local anesthetic from the intrathecal solution does not cause withdrawal, mortality or serious adverse events
Arm/Group | Bupivacaine + Opioid | Opioid
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 3/16 | 3/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bupivacaine + Opioid (N=16) | Opioid (N=16)
headache (Nervous system disorders) | 3 | 1
numbness/tingling (Nervous system disorders) | 1 | 2
nausea (Nervous system disorders) | 2 | 1
fatigue (General disorders) | 0 | 1
anxiety (Psychiatric disorders) | 0 | 1
skin irritation (Skin and subcutaneous tissue disorders) | 0 | 1
urinary hesitancy (Renal and urinary disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2016-01-29): https://cdn.clinicaltrials.gov/large-docs/86/NCT02886286/Prot_SAP_ICF_000.pdf